CLINICAL TRIAL: NCT06818019
Title: WIthdrawal of DUpilumab in Severe Asthma: a Randomized Non-inferiority-controlled Trial
Brief Title: Withdrawal of Dupilumab in Severe Asthma
Acronym: WIDUSA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/24/0325; 2024-516789-13-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-19; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Severe Asthma
Keywords: severe asthma; dupilumab; exacerbation; discontinuation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Multicentre open-label non-inferiority randomised controlled trial with two parallel groups, ratio 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stopping dupilumab (Experimental): The experimental strategy comprises stopping dupilumab with no dose-reducing or interval of time-increasing strategy from the day of inclusion/randomisation
  Interventions: Drug: Stopping dupilumab
- Dupilumab continuation (No Intervention): Dupilumab continuation at the same dose and same interval as baseline

INTERVENTIONS:
Drug: Stopping dupilumab — Stopping dupilumab with no dose-reducing or interval of time-increasing strategy
  Arms: Stopping dupilumab

SUMMARY:
Asthma management has been revolutionised by the development of biological therapies. Dupilumab is an anti-interleukin4 receptor marketed in 2020 for severe asthmatic patients with 2 exacerbations or more within the last 12 months. Although data showed that safety and efficacy of dupilumab are sustained when treatment is extended up to 3 years, no study has emerged regarding dupilumab discontinuation. This study aims to demonstrate the non-inferiority regarding strategy failure at 24 months of stopping dupilumab (intervention group) compared with its continuation (control group) in controlled asthma patients receiving this drug for at least 3 years.

DETAILED DESCRIPTION:
Although dupilumab is a very effective drug in severe asthma, the optimal duration of this drug is unknown. However, this is a crucial question given the high cost of dupilumab and the lack of data regarding the long-term inhibition of type 2 pathway. Studies on biologic discontinuation are scarce in severe asthma. Studies with other biologics have shown that discontinuation of these drugs is feasible particularly for patients with low exacerbation rate before stopping treatment. In a study with pooled asthma biologics, 1247 (25.1%) stopped the biologic among the 4958 biologic users (including 19.8% of dupilumab users). Among all stoppers, 10.2% failed discontinuation of the asthma biologic in the 6 months after stopping, defined as an increase of 50% or more in exacerbations. Among patients who continued the biologic, 9.5% had an increase of 50% or more in exacerbations during a 6-month period, showing a similar failing rate. Such data for dupilumab discontinuation are lacking.

In this study, we plan to include patients with controlled asthma treated with dupilumab for at least 3 years who will be randomised to stopping dupilumab or dupilumab continuation with a follow-up of 24 months.

In total, 5 visits will occur for each patient: the inclusion/randomisation visit (baseline), 3 follow-up visits at month 6, month 12, month 24 as usually done in severe asthma, and a phone call visit at 18 months for exacerbations, treatments and adverse events collection. At each onsite visit, asthma medications, concomitant treatments, nasal polyp score (if applicable), number of exacerbations, Asthma Control Questionnaire, Severe Asthma Questionnaire, Treatment Burden Questionnaire and Sino-Nasal Outcome Test-22 scores, Forced expiratory volume in one second, Forced vital capacity, Fraction exhaled nitric oxide (if available), blood eosinophil, neutrophil and lymphocyte counts, adverse events, hospital admissions, and unscheduled medical visits will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old
* Treated with dupilumab for at least 36 months for severe asthma
* Well controlled asthma defined by an Asthma Control Questionnaire score ≥ 18 and 0 or 1 exacerbation within the year prior to the inclusion visit

Exclusion Criteria:

* Patients who refuse to discontinue dupilumab, for any reason
* Patients with Forced expiratory volume in one second ≤ 30% of predicted values
* Patients treated by an oral corticosteroid dose ≥ 10 mg/day (in prednisone equivalent)
* Patients who have to discontinue dupilumab for a reason other than controlled asthma, such as an adverse drug reaction, a planned or current pregnancy, or a planned switch to another biologic indicated in severe asthma
* Patients who have to continue dupilumab for the treatment of comorbidities apart from nasal polyposis
* Active smoking
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2025-04-02 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Strategy failure | 24 months
  Proportion of patients with strategy failure defined as patients with an annualised number of asthma exacerbations ≥ 2 and/or dupilumab resume or switch to another biologic within 24 months following randomisation

SECONDARY OUTCOMES:
Change in asthma control test score | 6, 12 and 24 months
  Comparing the interventional group with the control group regarding the change in asthma control test score at 6, 12 and 24 months compared to baseline. The asthma control test score is a self-administered questionnaire consisting of 5 questions related to the frequency of asthma symptoms and the use of rescue treatments over the past 4 weeks. The score ranges from 5 (poorest control) to 25 (perfect control)
Resumption of dupilumab | 6, 12 and 24 months
  Proportion of patients with resumption of dupilumab in the interventional group (stopping dupilumab) at 6, 12 and 24 months
Adverse events or serious adverse events | 24 months
  Proportion of patients with adverse events or serious adverse events in both groups
Time to loss of control | 24 months
  Comparing the interventional group with the control group regarding the time between baseline to loss of control defined by a reduction of 5 points or more on asthma test control score
First exacerbation | 24 months
  Comparing the interventional group with the control group regarding the time to first exacerbation
Number of exacerbations | 24 months
  Comparing the interventional group with the control group regarding the number of exacerbations within 24 months
Proportion of patients with ≥ 1 exacerbation(s) | 6, 12 and 24 months
  Comparing the interventional group with the control group regarding the proportion of patients with ≥ 1 exacerbation(s) or severe exacerbation(s) at 6, 12 and 24 months. A severe exacerbation is defined as an emergency room visit or hospital admission or death related to asthma exacerbation.
Change in quality of life | 6, 12 and 24 months
  Comparing the interventional group with the control group regarding the change in quality of life at 6, 12 and 24 months compared to baseline.
  The change in the severe asthma questionnary quality of life score and the Burden of Treatment Questionnaire score at 6, 12 and 24 months compared to baseline.
  The severe asthma questionnary is a health-related quality of life questionnaire validated for use in severe asthma. It is scored using the mean value of 16 items (severe asthma questionnary score) in addition to a single item global rating of health-related quality of life. The Burden of Treatment Questionnaire is a 15-item questionnaire that assesses the treatment burden of chronic diseases.
Change in lung function | 6, 12 and 24 months
  The lung function change is a qualitative clinical criteria of failure/success of the strategy. This failure is made up of 3 components : Forced Expiratory Volume in 1 second (in L and % predicted, pre- and post-bronchodilator), Forced Vital Capacity (in L and % predicted) and forced exhaled nitric oxide (in ppb) at 6, 12 and 24 months compared to baseline
Change in the daily dose of oral corticosteroids | 6, 12 and 24 months
  Comparing the interventional group with the control group regarding the change in the daily dose (mg/day) of oral corticosteroids (in prednisone equivalent) at 6, 12 and 24 months compared to baseline
Change in the daily dose of inhaled corticosteroids | 6, 12 and 24 months
  Comparing the interventional group with the control group regarding the change in the daily dose (μg/day) of inhaled corticosteroids (in beclomethasone equivalent) at 6, 12 and 24 months
Effect on nasal polyposis | 6, 12 and 24 months
  Comparing the interventional group with the control group regarding the change in nasal polyposis endoscopic score (if available) and Sino-Nasal Outcome Test-22 score at 6, 12 and 24 months compared to baseline.
  The french version of Sino-Nasal Outcome Test-22 is a further modification of the Sino-Nasal Outcome Test-20, a fully validated and easy-to-use outcome measure in rhinology. In addition to the normal 20-item version of the Sino-Nasal Outcome Test, 2 additional items were measured, nasal blockage, and loss of sense of taste and smell. The 22-question Sino-Nasal Outcome Test-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent GUILLEMINAULT, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (29):
- France (29):
  - CHU de Toulouse, Toulouse, CHU de Toulouse
  - CHU Amiens-Picardie, Amiens, France
  - CHR d'Angers, Angers, France
  - CH de Bayonne, Bayonne, France
  - CHU de Besançon, Besançon, France
  - CHU de Brest, Brest, France
  - CHU de Caen, Caen, France
  - CH de Cannes, Cannes, France
  - CHU de Clermont-Ferrand, Clermont-Ferrand, France
  - CHI de Créteil, Créteil, France
  - CHU de Dijon, Dijon, France
  - CH Annecy Genevois, Epagny-Metz-Annecy, France
  - CHU Grenoble-Alpes, La Tronche, France
  - Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre, France
  - CH Le Mans, Le Mans, France
  - Institut Coeur Poumon, CHU de Lille, Lille, France
  - Hôpital Croix Rousse, Lyon, France
  - Hôpital Avicenne, Paris, France
  - Hôpital Européen Georges Pompidou, Paris, France
  - Hôpital Bichât, Paris, France
  - CHU de Bordeaux, Pessac, France
  - Hôpital Lyon Sud, Pierre-Bénite, France
  - CHU de Guadeloupe, Pointe à Pitre, France
  - CHU de Reims, Reims, France
  - CH de Roubaix, Roubaix, France
  - CHU de Nantes, Saint-Herblain, France
  - Nouvel Hôpital Civil, Strasbourg, France
  - Hôpital Foch, Suresnes, France
  - Hôpital Tarbes Lourdes, Tarbes, France